CLINICAL TRIAL: NCT03723954
Title: Evaluation of Heart Rate Variations of Golf Fans During the 2018 Edition of the Ryder Cup : the Ryder Heart Study
Brief Title: Heart Rate Variations of Golf Fans During the 2018 the Ryder Cup
Acronym: RyderHeart
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry); Boston Pharmaceuticals (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18_RIPH3-03
Record Dates: First submitted 2018-10-22; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Heart Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ECG Holter SpiderFlash-t — Record at visit V0 (day without match) and the competition days (Visit V1, V2 et V3) during the matches the heart rate of the golf fans.
  SpiderFlash-t™ from MicroPort is a long-lasting event recorder set in walking position by the investigator the day of the record and it is activated by detecting rhythm anomalies. This recorder is a Class IIA medical device (according to European Economic Community Directive 93/42). It benefits from European Economic marking.
Device: Actigraph GT3Xp — Record the study participant's physical activity while we record his heart rate.
  The GT3Xp based activity monitors provide objective measurements of human activity and are used in many research and clinical applications. It includes a micro-electro-mechanical system (MEMS) based accelerometer and an ambient light sensor. It benefits from CE marking and FDA agreement (Class II medical device).

SUMMARY:
Ryder Heart is an exploratory study of the heart rate variations of golf fans during the 2018 edition of the Ryder Cup. The main objective is to evaluate the impact of stress and strong emotions on heart rate variations and the occurrence of rhythmic anomalies in golf fans during this high-level golf competition. Such data are actually poorly described in medical and scientific literature.

DETAILED DESCRIPTION:
In 1996, a Dutch research team highlighted, for the first time, a strong statistical relationship between the outcome of a football match and cardiovascular mortality in men over 45 years of age. An excess mortality was reported among football fans on June 22nd 1996, day of the elimination of the Dutch by the French team during the penalty shoot-out of the European Champions League. A more recent study by Ute Wilbert-Lampen et al., confirmed the relationship between football matches of the 2006 World Cup and the occurrence of cardiovascular events such as rhythm disorders and coronary syndromes among football fans. Two factors favoring increased cardiovascular risk appear to emerge from these different studies: high-level football matches (most often played at home) and strong support and passion for one's sports team. However, the physiopathological mechanisms involved have not been fully understood yet. In addition, very little data exists on sports other than football. The investigators research hypothesis is that cardiovascular events induced by the passion of a sports fan could not be unique to only one sport. The Ryder Cup, one of the biggest sporting events in the world, is the ideal event to collect consolidation elements for the investigators hypothesis.

The main phase of the Ryder Heart study will take place during the Ryder Cup from the 28th till the 30th of September 2018.

ELIGIBILITY:
Inclusion Criteria:

* Man or a Woman golf fan ;
* At least 18 years old ;
* Either a healthy study volunteer or a study volunteer suffering from a heart disease ;
* With or without an implantable cardioverter-defibrillator ;
* Presence at the Golf National during at least one day of the Ryder Cup (September 28th and/or September 29th and/or September 30th, 2018);
* Presence and available for study inclusion :
* In the Ile de France zone on the eve of competition (September 27th, 2018);
* At Golf National at least two hours before matches' beginning at competition days ;
* In possession of official tickets issued by the organizers ;
* To accept to wear an ECG Holter for heart rate recording at inclusion (V0) and at least one competition day (from September 28th to September 30th, 2018).

Exclusion Criteria:

* Pregnant or lactating woman;
* Medical contraindication to ECG Holter ;
* Equipped with an implantable pacemaker ;
* Total dependence to stimulation of cardiac defibrillator;
* Suffering from a decompensated heart disease ;
* History of severe allergy to angioedema-type electrodes ;
* Body temperature under 36 celsius degree or equal or higher than 39 celsius degree at inclusion;
* Not opposed to the use of data collected via recording and electromagnetic measurements of heart rate (ECG) for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Golf fans attending at least one Ryder Cup match
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Record and measure by Spider Flash-t of the increase in the heart rate peak | 3 days
  The measure of the increase in the heart rate peak (in beats per minute) of study subjects at the days and times of golf matches will be performed with Spider Flash-t.
  The algorithms built into SpiderFlash-t detect episodes palpitations, syncope, atrial fibrillation and atrial flutter in addition to all other arrhythmias such as bradycardia and tachycardia in patients symptomatic and asymptomatic. The integrated SpiderFlash-t software includes a dedicated and specific algorithm for detect atrial fibrillation. This atrial fibrillation algorithm is independent of the algorithm main arrhythmia detection, also incorporated into SpiderFlash-t.
  So comparing the data recorded at V0 (baseline) with the data recorded during the golf match, a minimum increase in the heart rate peak of at least 10% (at days and times of golf meetings) will be considered a significant variation.

SECONDARY OUTCOMES:
average hourly variations of parameters related with heart rate | 3 days
  The exploratory nature of the Ryder Heart study does not allow adequate consideration of potential confounding factors that may affect heart rate. Thus, the variations of this heart rate can be described according to several characteristics: the intensity of the physical activity of the fans during the Ryder Cup using an Actigraph GT3Xp and the passion supporter for golf The data recorded by SpiderFlash-t will be analyzed by the analysis program of MicroPort. This program produces an automatic report of a classical and spectral analysis of the variability of the heart rate. The heart rate, its variability as well as the rhythmic events will thus be studied, with the description of the amplitudes, temporal, frequency and rhythmic parameters.
Fan's passion score for golf | 15 minutes
  The golf fan's degree of passion will be evaluated by a questionnaire including a series of items, inspired by studies by Vallerand et al. and Wann and Branscombe which help to classify the fans in three categories : little, moderately and very passionate.The scale includes 16 questions with answers choice going from 0 to 3. To whom will obtain a total score 0-16 = little passionate. To whom will obtain a total score 17-32 = moderately passionate. To whom will obtain a total score 33-48 = very passionate.
Record and measure fan physical activity by ActiGraph GT3Xp | 3 days
  The physical activity level of study participants will be quantified directly every day of competition, using a physical activity monitor / accelerometer type ActiGraph GT3Xp. This device will collect various information such as mouvements, gross acceleration, caloric flow, energy expenditure, active energy expenditure, the duration of physical activity and the number of steps of the supporter. The number of steps of the supporter is used to take into account a confounding factor (effect of the physical activity of the supporter on his heart rate) and estimate the main judgment criterion reliably.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DEMONIERE, MD, Principal Investigator — CHU deMartinique
Locations (1):
- Golf National, Saint-Quentin-en-Yvelines, France

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the main publication of the results, for not limited time.
Access Criteria: The conditions for the transfer of all or part of the database of the research are decided by the principal investigator / sponsor of the research and are the subject of a written contract.

REFERENCES:
- [Result] Spitters CE. Cardiovascular events during World Cup soccer. N Engl J Med. 2008 May 29;358(22):2408; author reply 2409. No abstract available. PMID 18512276
- [Result] Vallerand RJ, Ntoumanis N, Philippe FL, Lavigne GL, Carbonneau N, Bonneville A, Lagace-Labonte C, Maliha G. On passion and sports fans: a look at football. J Sports Sci. 2008 Oct;26(12):1279-93. doi: 10.1080/02640410802123185. PMID 18803066